CLINICAL TRIAL: NCT05849272
Title: Efficacy and Safety of Toluedesvenlafaxine Hydrochloride Extended-release Tablets in Somatic Symptoms of Depression: a Prospective, Single-arm, Multicenter Study
Brief Title: Efficacy and Safety of Toluedesvenlafaxine Hydrochloride Extended-release Tablets in Somatic Symptoms of Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMHC-DSS-001
Record Dates: First submitted 2023-04-23; First posted 2023-05-08 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Somatic Symptom
Keywords: medical treatment; somatic symptom; depression
MeSH Terms: conditions — Medically Unexplained Symptoms; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toludesvenlafaxine hydrochloride sustained-release tablets 80-160 mg group (Experimental): orally once a day
  Interventions: Drug: toludesvenlafaxine hydrochloride sustained-release tablets

INTERVENTIONS:
Drug: toludesvenlafaxine hydrochloride sustained-release tablets — orally once a day

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of toludesvenlafaxine hydrochloride sustained-release tablets in the treatment of somatic symptoms in depression, to provide evidence-based basis for clinical rational drug use.

DETAILED DESCRIPTION:
The study included 60 patients (aged 18 to 65 years) who meet the diagnostic criteria for depression in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and who are accompanied by physical symptoms.

All enrolled subjects were given toludesvenlafaxine hydrochloride sustained-release tablets monotherapy for 8 weeks, followed up at period of enrollment as baseline and at the end of 2th, 4th and 8th weeks. Adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects meet the Diagnostic and Statistical Manual of Manual Disorders, fifth Edition (DSM-5) criteria for depression;
2. Male or female aged ≥18 and ≤65 years;
3. Subject has a Hamilton Depression Rating Scale (HAMD-17) total score >17, anxiety/somatization factor ≥ 3;
4. Subject has a total score of Patient Health Questionnaire-15 (PHQ-15) ≥5;
5. Subject has a clear consciousness, no serious intellectual impairment, ability to speak autonomously, and no obvious symptoms of dementia;
6. Subjects voluntarily participate in the study and sign the informed consent form

Exclusion Criteria:

1. Allergic or known to be allergic to venlafaxine and desvenlafaxine;
2. Subjects whose previous treatment with venlafaxine have failed, or whose previous treatment with at least 2 different types of antidepressants are ineffective;
3. Subjects meet the diagnostic criteria for other psychotic disorders (except for depression) in DSM-5, personality disorders or intellectual disability, substance disorders or drug abuse within previous 6 months;
4. Subjects meet the diagnostic criteria for clinically significant unstable diseases, such as hepatic insufficiency or renal insufficiency, or cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatic, immune, infectious, skin and subcutaneous tissue diseases or metabolic disorders;
5. Subject has a severe self-injury/clear suicide attempt or behavior;
6. With blood pressure > 140/90 mmHg
7. Total bilirubin (TBIL) values 1.5 times / alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 2 times / creatinine (Cr) 1.2 times higher than the upper limit of normal, or Thyroid-stimulating hormone (TSH) outside the normal range at screening;
8. Electrocardiogram (ECG) abnormalities that are clinically significant at period of screening and that the investigator considers as inappropriate conditions for inclusion, such as QTc interval > 470 ms in men and QTc interval > 480 ms in female;
9. Subject has a history of moderate or severe brain trauma (for example, loss of consciousness ≥1 hour) or other neurological disorders or systemic diseases, which may affect the neurological function of CNS;
10. Pregnant or lactating women, recent planned pregnancy and unable to ensure effective contraception during the period;
11. Other conditions that the investigator considers the participant is not suitable for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-15 (PHQ-15) | 8 Weeks
  The PHQ-15 has a 15-item checklist. Items are rated on a scale of 0-2, for a total score range of 0 -30 (scores ≥ 5, ≥10, ≥15 represent mild, moderate and severe levels of somatization).
The Chinese version of the Somatization Symptom Scale (SSS-CN) | 8 Weeks
  The SSS-CN has a 20-item checklist. Items are rated on a scale of 1-4, for a total score range of 20-80 (scores between 20-29, 30-39, 40-59, ≥60 correspond normal, mild, moderate and severe levels of somatic symptom disorder).

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 8 Weeks
  The VAS is a validated, subjective measure for acute and chronic pain. The total score range of 0 -10 (from no pain to worst pain).
Multidimensional Fatigue Index (MFI-20) | 8 Weeks
  The MFI-20 has a 20-item checklist, consist of 5 subscales. Items are rated on a scale of 1-5, for a total score range of 20 -100 (high scores represent more fatigue) and each subscale range of 4-20.
Sheehan Disability Scale (SDS) | 8 Weeks
  The SDS has a 5-item checklist. The total scores range of 0 -30 (from no impairment to highly impairment of function of normal life).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, He M, Zhang H, Luo Y, Sun X, Yao Z, Tang H, Yan R, Du X, Li Z, Peng D, Wang Z. Efficacy and Safety of Toludesvenlafaxine Hydrochloride Sustained-Release Tablets on Somatic Symptoms of Major Depressive Disorder: A Prospective, Single-Arm, Multicenter Clinical Study. Neuropsychiatr Dis Treat. 2025 Jul 9;21:1387-1397. doi: 10.2147/NDT.S513481. eCollection 2025. PMID 40661857